CLINICAL TRIAL: NCT05910151
Title: Introduction of Tandem Mass Spectrometry (MS/MS) Technology in the Program of Selective Screening of Hereditary Metabolic Diseases in Kazakhstan
Brief Title: Selective Screening of Children for Hereditary Metabolic Diseases by Tandem Mass Spectrometry in Kazakhstan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West Kazakhstan Medical University (Other)
Responsible Party: Principal Investigator, Zharmakhanova Gulmira, Head of Department of Natural Sciences disciplines (with course of Molecular Biology and Medical Genetic), West Kazakhstan Medical University
Other Study IDs: IRN AP148699996
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Propionic/Methylmalonic Acidemias; Maple Syrup Urine Disease; Citrullinemia; Argininosuccinic Aciduria; Ornithine Transcarbamylase Deficiency; Carbamoyl Phosphate Synthetase I Deficiency; N-acetylglutamate Synthase Deficiency; Nonketotic Hyperglycinemia; Tyrosinemia; Homocystinuria; Arginase Deficiency; Isovaleric Acidemia; Short/Branched Chain Acyl-CoA Dehydrogenase Deficiency; Isobutyryl-CoA Dehydrogenase Deficiency; Glutaric Acidemia Type I; 3-methylcrotonyl-CoA Carboxylase Deficiency; Biotinidase Deficiency; Malonyl-CoA Decarboxylase Deficiency; Beta-ketothiolase Deficiency; 3-hydroxy-3-methylglutaryl-CoA Lyase Deficiency; 3-methylglutaconyl-CoA Hydratase Deficiency; Medium-chain Acyl-CoA Dehydrogenase Deficiency; Very Long-chain Acyl-CoA Dehydrogenase Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; Glutaric Acidemia Type II; Primary Carnitine Deficiency; Carnitine Palmitoyltransferase I Deficiency; Carnitine Palmitoyltransferase II Deficiency; Carnitine-acylcarnitine Translocase Deficiency
Keywords: Inborn errors of metabolism, MS/MS, selective screening
MeSH Terms: conditions — Maple Syrup Urine Disease; Citrullinemia; Argininosuccinic Aciduria; Ornithine Carbamoyltransferase Deficiency Disease; Carbamoyl-Phosphate Synthase I Deficiency Disease; N-acetyl glutamate synthetase deficiency; Hyperglycinemia, Nonketotic; Tyrosinemias; Homocystinuria; Hyperargininemia; Acidemia, isovaleric; 2-Methylbutyryl-CoA Dehydrogenase Deficiency; Isobutyryl-CoA dehydrogenase deficiency; Glutaric Acidemia I; 3-methylcrotonyl CoA carboxylase 1 deficiency; Biotinidase Deficiency; Malonic aciduria; Beta ketothiolase deficiency; 3-Hydroxy-3-Methylglutaryl-CoA Lyase Deficiency; 3-Methylglutaconic Aciduria, Type I; Medium chain acyl CoA dehydrogenase deficiency; VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Systemic carnitine deficiency; Carnitine palmitoyl transferase 1A deficiency; Carnitine palmitoyl transferase 2 deficiency; Carnitine-Acylcarnitine Translocase Deficiency; Metabolism, Inborn Errors | interventions — Aging

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2250 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- reference group A: healthy newborns aged 1-7 days
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From Healthy Newborns (Aged 1-7 Days)
- reference group B: healthy children aged 8 days - 7 years
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From Healthy Children Aged 8 Days - 7 Years
- reference group C: healthy children aged 8 - 18 years
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From Healthy Children Aged 8-18 Years
- selective group A: children aged 1 day - 7 days suspected with IEM
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From High-risk Newborns (Aged 1-7 Days)
- Selective group B: children aged 8 days - 7 years suspected with IEM
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From High-risk childrens (Aged 8 Days- 7 years)
- Selective group C: children aged 8-18 years suspected with IEM
  Interventions: Diagnostic Test: Obtaining Dry Blood Spots From High-risk childrens (Aged 8 - 18 years)

INTERVENTIONS:
Diagnostic Test: Obtaining Dry Blood Spots From Healthy Newborns (Aged 1-7 Days) — Neonatal blood samples will be taken from healthy infants no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs) for LC-MS/MS analysis. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers until analyzed by LC-MS/MS in accordance with standards from the Institute of Clinical and Laboratory Standards.
  Groups: reference group A
Diagnostic Test: Obtaining Dry Blood Spots From Healthy Children Aged 8 Days - 7 Years — Blood samples will be taken from healthy childrens no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs) for LC-MS/MS analysis. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers until analyzed by LC-MS/MS in accordance with standards from the Institute of Clinical and Laboratory Standards
  Groups: reference group B
Diagnostic Test: Obtaining Dry Blood Spots From Healthy Children Aged 8-18 Years — Blood samples will be taken from healthy childrens no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs) for LC-MS/MS analysis. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers until analyzed by LC-MS/MS in accordance with standards from the Institute of Clinical and Laboratory Standards
  Groups: reference group C
Diagnostic Test: Obtaining Dry Blood Spots From High-risk Newborns (Aged 1-7 Days) — Blood samples will be taken from high-risk infants no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs). The sample must be taken before transfusion therapy (or blood is taken no earlier than 48-72 hours after the transfusion) or extracorporeal membrane oxygenation. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers.
  Groups: selective group A
Diagnostic Test: Obtaining Dry Blood Spots From High-risk childrens (Aged 8 Days- 7 years) — Blood samples will be taken from high-risk childrens no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs). The sample must be taken before transfusion therapy (or blood is taken no earlier than 48-72 hours after the transfusion) or extracorporeal membrane oxygenation. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers
  Groups: Selective group B
Diagnostic Test: Obtaining Dry Blood Spots From High-risk childrens (Aged 8 - 18 years) — Blood samples will be taken from high-risk childrens no earlier than 3 hours after feeding by heel prick with a heel stick. Five drops of whole blood (~75 µl each) will be applied to Guthrie cards, Ahlstrom 226 filter paper, PerkinElmer 226 Five-Spot Card (PerkinElmer Health Sciences, Greenville, USA) to form dried blood spots (DBSs). The sample must be taken before transfusion therapy (or blood is taken no earlier than 48-72 hours after the transfusion) or extracorporeal membrane oxygenation. Samples will be dried for 4 hours at room temperature and then stored at 4°C in individually labeled zippered plastic bags with desiccants or other sealed containers
  Groups: Selective group C

SUMMARY:
Inborn errors of metabolism (IEM) are not have specific clinical signs, they masquerade as other diseases, and are difficult to diagnose using only clinical manifestations or routine laboratory tests. IEM most commonly manifest in early infancy and childhood. Despite the fact that most IEM are rare in the population, they occupy one of the first places in the structure of childhood pathology, early infant mortality and disability. IEM often remains undiagnosed, while timely diagnosis and timely treatment started can prevent severe systemic damage leading to death and disability. The appointment of a special treatment (diet therapy, cofactors, enzyme replacement therapy) prevents or significantly inhibits the development of the pathological process, especially if the diagnosis is made in the early stages of the disease. To start pathogenetic treatment as early as possible, it is necessary to diagnose IEM as accurately and as early as possible.

Among the diseases included in mass screening programs IEM are especially important due to the development of disability and early mortality in the absence of timely diagnosis and treatment, as well as a high risk of recurrence in burdened families. In this connection, the main goals of mass screening - the prevention of disability in children and the reduction of early infant mortality - dictate the need to introduce modern technologies for preclinical diagnosis of IEM.

Based on the results of the study, it is planned to scientifically substantiate the need for the introduction of selective screening of children for hereditary metabolic diseases using the technology of tandem mass spectrometry in the Republic of Kazakhstan for timely diagnosis, therapy of IEM and prevention of disability. The introduction of a selective newborn screening program for IEM should always be preceded by a study aimed at studying the prevalence of the disease in a certain region, determining regional reference values of the studied metabolites. Local incidence and outcome data can be used to persuade health officials to prioritize screening in health care spending.

The main scientific question and hypothesis of the project is whether it is necessary to introduce tandem mass spectrometry technology in the neonatal screening program for IEM.

DETAILED DESCRIPTION:
In Kazakhstan, the use of MS/MS in metabolic screening programs is in development. This is due to the high cost of equipment and consumables, as well as the lack of special screening centers and specialists.

Selective screening is an important tool for diagnosing various types of inborn errors of metabolism (IEM). Currently, MS/MS-based technologies are widely used, which allow the simultaneous determination of the amount of several metabolites (amino acids, acylcarnitines) from a very small amount of a biological sample. However, age reference cutoff ranges for each analyte should be established first for each population prior to screening as cutoffs depend on various factors such as genetic background, population geographic location, diet, sex, age.

Data on the prevalence of most IEMs, with the exception of phenylketonuria, are not available in Kazakhstan. The data obtained in this study will make it possible to conduct a comparative analysis of the prevalence of IEM in Asia and establish reference values for the concentrations of amino acids and acylcarnitines in the blood of newborns for the Kazakhstan population. Newborn sreening is currently being conducted in Kazakhstan for two hereditary diseases - phenylketonuria and congenital hypothyroidism, which are the most represented screening diseases in most countries. A nationwide newborn screening program for two mandatory diseases, congenital hypothyroidism and phenylketonuria (PKU), began in 2007. ENBS on aminoacid disorders (AAD), organic acidemias (OA) and fatty acid oxidation defects (FAOD) is not conducted in Kazakhstan.

For Kazakhstan, as a country that does not have a mandatory ENBS program, selective screening can be an important tool for diagnosing IEM. The present study aims to develop and validate an MS/MS method for the simultaneous determination of 51 metabolites in DBS for IEM screening, as well as the determination of age-related amino acid ranges, acylcarnitines and succinylacetone in children's population of Kazakhstan. Our selective screening was initiated to obtain data on the incidence of IEM in children at risk in Western Kazakhstan. From October 2022 to December 2024, the frequency of 37 AAD, OA and FAOD will be assessed using LC-MS/MS technology in a group of children at high risk. A summary report will be presented on the screening of high-risk children for IEM in Western Kazakhstan using the LC-MS/MS method.

The results of selective screening tests in different age groups of subjects should be interpreted by comparison with the reference values and/or cut-off levels established for these groups. It is generally accepted that children need to use reference populations that reflect changes associated with growth and development. Therefore, one of the objectives of this study is to establish reference intervals for the concentration of amino acids and acylcarnitines in dry blood spots for different age groups in the range from 1 day to 18 years.

The goal of this observational study is to сonduct selective screening for IEM among children of Kazakhstan aged from 1 day to 18 years using tandem mass spectrometry to determine the prevalence of IEM and reference values of metabolites followed by subsequent substantiation of the need to introduce selective screening of newborns for IEM by MS/MS.

The main questions it aims to answer are:

question 1: what are the reference values of metabolites (amino acids and acylcarnitines) in different age groups of children in Kazakhstan; question 2: what is the contribution of IEM to the structure of the pathology of the nervous system in young children and is it necessary to introduce tandem mass spectrometry technology in the neonatal screening program for IEM?

ELIGIBILITY:
Inclusion Criteria:

Referense group: Healthy male and female children aged 1 day to 18 years. Newborns born during the study period (all newborns will be included in this study will meet all selected inclusion criteria to ensure that they do not suffer from any disorder or disease. Healthy male and female newborns must weigh within 2500 -4000 g, gestational age 37-42 weeks, Apgar score above 7 for 10 min.) Sample group: children aged 1 day to 18 years will be selected if one of the main criteria or two or more additional criteria (symptoms) is identified.

Main criteria (symptoms): 1) Sudden deterioration in the clinical condition of the child after a period of normal development (days, weeks, months): acute metabolic encephalopathy, lethargy (coma), seizures resistant to antiepileptic therapy. 2) Hepatomegaly (hepatosplenomegaly). 3) Metabolic acidosis with an increase in the anion gap. 4) Multiple fractures. 5) Child mortality in the family from diseases with similar symptoms.

Additional criteria (symptoms): Treatment-resistant seizures; Abnormal muscle tone: dystonia, hyperkinesis, hypotension; Speech delay; Mental retardation of unknown cause; Cardiomyopathy; Tachypnoea; Frequent spitting up (vomiting); Osteo-articular abnormalities (joint stiffness, chest deformity, rickets-like changes); Hernias (umbilical, inguinal-scrotal); Persistent or recurrent hypoglycemia; Metabolic alkalosis; Increase in ketone bodies in the blood and (or) urine; Hyperammonemia; Increase in the level of liver enzymes (AlAT, AST) more than 1.5 times the norm; Increase in the level of creatine phosphokinase (CPK) more than 2 times the norm; Decrease in the level of alkaline phosphatase (AP) below the age norm; Imaging or electrophysiological studies suggesting metabolic disorders; Leukopenia; Thrombocytopenia; Abnormal urine, body, ear wax, any unusual smell; Hair growth disorders, alopecia; Ophthalmological anomalies; Unusual appearance, dysmorphic features; History of previous sibling death of unknown cause; Parents' consanguinity; A positive family history of metabolic disorders.

Exclusion Criteria:

The study will exclude patients who has:

1. perinatal brain injury,
2. brain injuries,
3. infections of the central nervous system,
4. toxicological diseases,
5. tumors,
6. chromosomal abnormalities,
7. with the symptoms specified in the inclusion criteria, but with a confirmed diagnosis of any disease other than amino acids disorders (AAD), fatty acid oxidation defects (FAOD) or organic academias (OA).

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: To establish reference values for metabolites, healthy participants without any disease will be included in the study: 750 healthy male and female children aged 1 day to 18 years old from West Kazakhstan will be recruited and included in the study. Depending on age, healthy children will be divided into the following groups: group A (age 1-7 days), group B (age 8 days-7 years) and group C (age 8-18 years).
  A total of 1,500 children from the West Kazakhstan population (age 1 days -18 years) with suspected metabolic disorders will be referred by primary care neonatologists and pediatric consultants based on their clinical symptoms associated with metabolic disorders and examined for IEM.
Sampling Method: Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of the concentration value of amino acids and acylcarninits activity in Dry blood spots among Newborns and Children in Kazakhstan | Two years
  Amino acids: Alanine (Ala), Arginine (Arg), Citrulline (Cit), Glutamine (Gln), Glutamic acid (Glu), Glycine (Gly), Leucine (Leu), Isoleucine (Leu), Hydroxyproline (Leu), Methionine (Met), Ornithine (Orn), Phenylalanine (Phe), Proline (Pro), Tyrosine (Tyr), Valine (Val). Acylcarninits: free carnitine (C0), Acetylcarnitine (C2), Propionylcarnitine (C3), Malonylcarnitine+3-Hydroxybutyrylcarnitine (C3DC/C4OH), Butyrylcarnitine (C4), Methylmalonylcarnitine+3-Hydroxyisovalerylcarnitine (C4DC/C5OH), Isovalerylcarnitine (C5), Tiglylcarnitine (C5:1), Glutarylcarnitine (C5DC), Hexanoylcarnitine (C6), Octanoylcarnitine (C8), Octenoylcarnitine (C8:1), Decanoylcarnitine (C10), Decenoylcarnitine (C10:1), Decadienoylcarnitine (C10:2), Dodecanoylcarnitine (C12), Hydroxydodecenoylcarnitine (C12:1), Myristoylcarnitine (C14), Tetradecenoylcarnitine (C14:1), Tetradecadienoyl-carnitine (C14:2), Hydroxytetradecanoylcarnitine (C14OH), Palmitoylcarnitine (C16), Hexadecenoylcarnitine (C16:1), Hydroxy-Hexad

CONTACTS AND LOCATIONS:
Overall Officials: Gulmira M. Zharmakhanova, MD, PhD, Principal Investigator — West Kazakhstan Medical University; Lyazzat M. Syrlybayeva, MD, Study Chair — West Kazakhstan Medical University; Victoria I. Kononets, MD, MS, Study Chair — West Kazakhstan Medical University
Locations (1):
- Regional perinatal center of Aktobe region, Aktobe, Aktobe Region, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zharmakhanova G, Kononets V, Balmagambetova S, Syrlybayeva L, Nurbaulina E, Zhussupova Z, Sakhanova S, Ayaganov D, Kim S, Zhumalina A. Selective screening for inborn errors of metabolism using tandem mass spectrometry in West Kazakhstan children: study protocol. Front Genet. 2024 Jan 12;14:1278750. doi: 10.3389/fgene.2023.1278750. eCollection 2023. PMID 38283151